CLINICAL TRIAL: NCT06952829
Title: Randomized Controlled Clinical Trial Assessing the Effectiveness of a Venipuncture Strategy Adapted According to A-DIVA Score Results Compared to Standard Care in Reducing the Number of Punctures
Brief Title: Evaluation of A-DIVA Score Effectiveness at Admission for Preserving Venous Capital in Patients With Difficult Access
Acronym: ERV-ADIVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Robert Ballanger (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GHT_CHIRB_20240618
Record Dates: First submitted 2025-02-04; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Internal Medicine; Surgery; Neurology
Keywords: Adult-Difficult IntraVenous Access (A-DIVA); capital venous preservation

STUDY DESIGN:
Intervention Model Description: controlled, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with Adult-Difficult IntraVenous Access (A-DIVA) and with A-DIVA modified score evaluation (Experimental): intravenous access of these patients will be evaluated by the ADIVA and with modified ADIVA (ADIVA m) scores before puncture by the nurse
  Interventions: Other: evaluation of intravenous access of patients with Adult-Difficult IntraVenous Access (A-DIVA) score prior to puncturing subject; Other: evaluation of intravenous access of patients with modified Adult-Difficult IntraVenous access(A-DIVA modified) score prior to puncturing subject
- without Adult-Difficult IntraVenous Access (A-DIVA) score evaluation (No Intervention): control group, patients will not undergo an evaluation of their intravenous access using the Adult-Difficult IntraVenous Access (A-DIVA) tool prior to peripheral IV catheter placement. They will receive standard care as routinely provided in the hospital.

INTERVENTIONS:
Other: evaluation of intravenous access of patients with Adult-Difficult IntraVenous Access (A-DIVA) score prior to puncturing subject — The patient's intravenous access will be evaluated using the A-DIVA score by the study nurse at the time of admission, prior to venipuncture performed by the care nurse
  Arms: with Adult-Difficult IntraVenous Access (A-DIVA) and with A-DIVA modified score evaluation
Other: evaluation of intravenous access of patients with modified Adult-Difficult IntraVenous access(A-DIVA modified) score prior to puncturing subject — The patient's intravenous access will be evaluated using the A-DIVA-m score by the study nurse at the time of admission, prior to venipuncture performed by the care nurse
  Arms: with Adult-Difficult IntraVenous Access (A-DIVA) and with A-DIVA modified score evaluation

SUMMARY:
In certain cases (e.g.: patient who are difficult to perfuse, thin veins, etc.), an increase in venipunctures performed by study nurses in healthcare services can lead to a loss of venous capital, repeated pain during punctures, discontinuous treatment follow-up and numerous requests for assistance from colleagues, including nurse anesthetists, but often too late.

The main objective of project is to reduce the number of punctures to access the venous system after evaluation of adult patients upon entering the hospitalization department using the A-DIVA tool. the A-DIVA score predicts the difficulty in infusing an adult patient

DETAILED DESCRIPTION:
This research evaluates the importance of assessing the venous capital access of hospitalized patients prior to the placement of an intravenous infusion, in order to save time in initiating therapeutic treatment and to prevent or reduce the number of venipunctures and the associated inconveniences (pain, discontinuous treatment monitoring). This approach aims to preserve the patient's venous capital.

In the proposed study, investigators will evaluate the patients' venous capital using the Adult-Difficult IntraVenous Access (A-DIVA) tool upon hospital admission and during hospitalization before any peripheral intravenous (IV) catheter placement.

During the inclusion visit, after obtaining informed consent, patients will be randomized into one of two groups:

* Group A: Patients will undergo an evaluation of their venous capital by a study nurse using the Adult-Difficult IntraVenous Access (A-DIVA) tool prior to any peripheral IV catheter placement during hospitalization.
* Group B: Patients will not undergo an evaluation of their venous capital using the Adult-Difficult IntraVenous Access (A-DIVA) tool prior to peripheral IV catheter placement. They will receive standard care as routinely provided in the hospital ward.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Adult Patients Aged 18 Years and Older
* written informed consent given by patient
* Affiliation to a social security system or equivalence system

Exclusion Criteria:

* Patients in Intensive Care Units
* Patients with Psychiatric Disorders or Under Psychiatric Care
* Minor Patients Under 18 Years of Age
* Pregnant or Breastfeeding Women
* Vulnerable and Protected Individuals as Defined by the Public Health Code (Articles L.1121-5 to L.1121-8 and L.1122-1-2)
* Patients Participating in Another Interventional Study
* Dying patients
* Patients Receiving Infusions of:

  * Chemotherapy Drugs with a pH <5 or >8
  * Solutions with an Osmolarity >900 mOsm/L
* Patients refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of Venipunctures Performed to Establish the First Peripheral Intravenous Line in the Hospital services | Periprocedural Venipuncture performed by study nurse from Day 0 (date of admission to hospital service) to Day 10 or until hospital discharge subject
  Number of Venipunctures Performed to Establish the First Peripheral Intravenous Line in the Hospital services

SECONDARY OUTCOMES:
pain score (numeric rating scale) during venipuncture | During venipuncture from Day 0 to Day 10 or throughout the entire hospitalization period
  assess the patient's pain on a scale of 0 to 10 at the time of the puncture. A lower score indicates less painful, a higher score means that patient is more painful.
duration of successful catheter placement | During catheter placement from Day 0 to Day 10 or throughout the entire hospitalization period
  duration of successful catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Eric MORTUREUX, IADE, Principal Investigator — CH BALLANGER
Locations (1):
- CHI Robert Ballanger, Aulnay-sous-Bois, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490
- [Background] Heydinger G, Shafy SZ, O'Connor C, Nafiu O, Tobias JD, Beltran RJ. Characterization of the Difficult Peripheral IV in the Perioperative Setting: A Prospective, Observational Study of Intravenous Access for Pediatric Patients Undergoing Anesthesia. Pediatric Health Med Ther. 2022 May 4;13:155-163. doi: 10.2147/PHMT.S358250. eCollection 2022. PMID 35548373
- [Background] van Loon FHJ, van Hooff LWE, de Boer HD, Koopman SSHA, Buise MP, Korsten HHM, Dierick-van Daele ATM, Bouwman ARA. The Modified A-DIVA Scale as a Predictive Tool for Prospective Identification of Adult Patients at Risk of a Difficult Intravenous Access: A Multicenter Validation Study. J Clin Med. 2019 Jan 26;8(2):144. doi: 10.3390/jcm8020144. PMID 30691137